CLINICAL TRIAL: NCT05802446
Title: Real-time fMRI Neurofeedback as Treatment for Inter-critical Mood Symptoms in Bipolar Disorder : a Randomized Controlled Multicentric Trial
Brief Title: Neurofeedback for Bipolar Disorder
Acronym: NEUROFEED-BD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP180597
Record Dates: First submitted 2023-02-28; First posted 2023-04-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Neurofeedback; fMRI; Residual symptoms; Emotion; Cognitive training
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active feedback (Experimental): Group receiving "real" neurofeedback (NFB) (activity of the emotional brain network)
  Interventions: Other: Real-time fMRI Neurofeedback
- Sham feedback (Sham Comparator): Group receiving "sham" NFB (activity from brain regions not implicated in emotion processing) to control for a potential placebo effect.
  Interventions: Other: Real-time fMRI Neurofeedback

INTERVENTIONS:
Other: Real-time fMRI Neurofeedback — Neurofeedback with real-time fMRI is a recent technique that allows to record the BOLD signal from a particular brain region and to display it back in real-time to the participant. With this feedback on brain activity, subjects can learn to control the activity of selected brain areas. Trial after trial, participants develop their individual strategies to voluntarily regulate the signal. The main objective of the neurofeedback training is that the participant develops an enhanced ability to exert control over activity in the target area(s) even without feedback. By manipulating targeted brain circuits, this training can induce modifications in particular behaviors and promote selective plasticity within the corresponding brain networks.

SUMMARY:
Bipolar Disorder (BD) is a severe mood disorder affecting between 1% and 3% of the general population. It is characterized by the succession of depressive and manic episodes, with periods of stabilization during which patients may present "residual" depressive or anxious symptoms, which are characterized by sadness and emotional hyper-reactivity. Although subthreshold, these residual symptoms are very disabling for their daily lives and are associated with the risk of recurrence and poor global functioning. The effect of pharmacological and psychotherapeutic treatments is demonstrated in the management of acute episodes but remains insufficient on residual symptoms. Therefore, there are so far few therapeutic options to target the inter-episode residual symptoms in BD. One novel approach is the real-time functional magnetic resonance imaging (fMRI) neurofeedback (NFB), which has already been shown to be an efficient method for self-regulating brain function, behavior and treating depression.

Hypothesis/Objective :

This study aims at assessing the efficacy of 3-weeks neurofeedback training with real-time fMRI on the treatment of residual mood symptoms in patients with BD. The investigators will specifically target depressive symptoms by training the patients to regulate the emotional network hemodynamic response to emotional stimuli.

Method :

The investigators will include 64 stabilized patients with BD. The investigators will recruit them in three French expert centers for BD and will randomly assign them to the experimental group, receiving feedback from the emotional brain network hemodynamic activity, or to the control group, receiving the signal from control brain areas not involved in emotion processing. Both groups will be trained to regulate their brain activity while they are presented with negatively valenced emotional pictures, based on the neurofeedback shown immediately after the trial. They will continue their usual treatment (as prescribed) throughout the duration of the study. Clinical scales and cognitive tests will enable us to evaluate the symptomatic, emotional, and cognitive changes after NFB training. The investigators will also measure resting-state functional connectivity and brain morphology before and after NFB to assess brain plasticity and to explore the neural mechanisms associated with successful regulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bipolar disorder I or II (DSM-5 criteria);
* Aged between ≥ 18 and ≤ 65;
* Absence of major mood episode for at least 3 months before inclusion (MADRS scores < 12; YMRS score < 10);
* Presence of residual depressive symptoms, as assessed by the MADRS (score > 5);
* Stabilized dose of mood stabilizer medication for at least 3 months before inclusion.
* Written consent
* Affiliation to a social security system
* Effective contraception for women of childbearing age

Exclusion Criteria:

* Severe physical disorders that may be life-threatening;
* Major psychiatric (Axis 1) comorbidities except for anxiety disorders;
* Any current substance abuse except for tobacco or cannabis. Substance abuse will be defined by the DSM V criteria;
* Exclusion criteria applicable to MRI Panic disorder, claustrophobia, epilepsy Pace maker or neuronal stimulator, intraocular or intracerebral metallic foreign body, cochlear implant, cardiac valve or metallic surgical arterial material, non removable removable magnetizable metallic material
* Somatic disorder that may affect cognitive abilities and brain structures (e.g., HIV infection, MS, lupus, Parkinson's disease, epilepsy, dementia...);
* Ongoing non-pharmacological treatment: structured psychotherapeutic interventions (Cognitive Behavioral Therapy - CBT, Interpersonal and Social Rhythm Therapy - IPSRT) as well as brain stimulation techniques (Electroconvulsive Therapy - ECT, Transcranial Magnetic Stimulation - TMS, Deep Brain Stimulation - DBS);
* Subject included in clinical and / or therapeutic experimentation in progress.
* Patients under legal protection
* Prisoners
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Baseline, 3 weeks.
  Evaluation of depressive symptoms. Total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms.

SECONDARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale (MADRS) | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of depressive symptoms. Total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms.
Young Mania Rating Scale (YMRS) | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of manic symptoms. Total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms.
Bipolar Depression Rating Scale (BDRS) | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of bipolar depression. Total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms.
State-Trait Anxiety Inventory (STAI A-B) | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of trait and state anxiety. Total score ranging from 20 to 80 for both subscales, with higher scores indicating a greater severity of symptoms.
Multidimensional Assessment of Thymic States - MAThyS | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of thymic state. Total score ranging from 0 to 200, lower scores indicate general inhibition, and higher scores indicate general excitation. A more descriptive approach can be done by analysing the sub-score.
Affective Intensity Measure - AIM | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of emotion reactivity. Total score ranging from 20 to 120, with higher scores indicating higher strength or intensity of people's emotional experiences.
Affective Lability Scale - ALS | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of mood lability. Total score ranging from 0 to 162, with higher scores indicating greater affective lability.
Cognitive Emotion Regulation Questionnaire - CERQ | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of emotion regulation abilities. Subscales scores ranging from 4 to 20, with higher subscale scores indicating greater use of a specific cognitive strategy.
Quality of life scale - QOLS | Baseline, 3 weeks, and 4, 8 weeks after the end of the training. .
  Quality of life assessment. Score ranging from 1 to 5, 5 indicating better quality of life
Five Facets Mindfulness Questionnaire - FFMQ | Baseline, 3 weeks and 4, 8 weeks after the end of the training.
  Evaluation of trait mindfulness. Total score ranging from 39 to 195, higher scores are indicative of someone who is more mindful in their everyday life
Global functioning assessment - GAF scale | Baseline, 3 weeks, and 4, 8 weeks after the end of the training.
  Evaluation of global functioning. Total score ranging from 0 to 100, higher scores indicating better global functioning.
Questionnaire of Adherence to the technology | Baseline, 3 weeks.
  Evaluation of the score of the acceptability of neurofeedback. Total score ranging from 6 to 42, higher scores indicating better acceptability of the technology.
Self-efficacy scale | Baseline, 3 weeks.
  Evaluation of personal efficiency. Total score ranging from 21 to 105, higher scores indicating stronger belief that one's actions are responsible for successful outcomes.
The Ekman facial recognition test | Baseline, 3 weeks.
  Emotion recognition evaluation. Cognitive task
The affective bias task | Baseline, 3 weeks.
  Evaluation of emotional bias. Cognitive task
The Test battery for Attentional Performance (TAP) | Baseline, 3 weeks.
  Evaluation of attention. Cognitive task
The choice reaction task | Baseline, 3 weeks.
  Evaluation of mindwandering, meta-awareness and ruminations. Cognitive task
MRI T1-T2 weighted scan | Baseline, 3 weeks
  Evaluation of grey and white matter (micro)structure. MRI measurement
MRI diffusion weighted scan | Baseline, 3 weeks
  Evaluation of grey and white matter (micro)structure. MRI measurement
functional MRI resting-state scan | Baseline, 3 weeks
  Evaluation of brain functional connectivity. MRI measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Chenevier, Créteil, val-de-marne, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION